CLINICAL TRIAL: NCT05564975
Title: Construction and Application of Pressure Injury Risk Prediction Model for Critically Ill Patients Based on Machine Learning Algorithm
Brief Title: Construction and Application of Pressure Injury Risk Prediction Model for Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yang Chaonan (Other)
Responsible Party: Sponsor-Investigator, Yang Chaonan, Nurse-in-charge, The First People's Hospital of Huzhou
Organization: The First People's Hospital of Huzhou (Other)
Other Study IDs: 2022KYLL053
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Pressure Injury; Critically Ill Patients; Risk Factors; Machine Learning Algorithms
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospital-acquired pressure injury group: According to the hospital adverse event management system, patients diagnosed with pressure injury in the hospital were included in the HAPI group, and patients who reported high risk of pressure injury during the same period were selected and included in the non-HAPI group.
- No-hospital-acquired pressure injury group: According to the hospital adverse event management system, patients diagnosed with pressure injury in the hospital were included in the HAPI group, and patients who reported high risk of pressure injury during the same period were selected and included in the non-HAPI group.

INTERVENTIONS:
Other:

SUMMARY:
In the previous investigation, investigators found that when the risk factors of stress injury in critical patients changed, clinical nurses lacked the awareness of evaluating the risk of stress injury, and lacked the risk assessment of this link. The stress risk prediction model is based on etiology. By analyzing the risk factors, the machine learning algorithm is used to evaluate the risk of pressure damage, and the prediction model of pressure damage can dynamically and comprehensively evaluate its risk. It is also a risk assessment tool. At present, there is no research on applying the stress injury risk prediction model of critical patients to the intensive care information software in China. In this study, the artificial intelligence algorithm library will be used to construct and apply the stress injury risk prediction model for critical patients.

DETAILED DESCRIPTION:
1.1 Epidemiological characteristics of hospital-acquired pressure injuries in critically ill patients As one of the global health problems, stress injury is a common problem faced by medical and health institutions, and it is considered as the most serious hospital-acquired adverse event. Hospital Acquired Pressure Injury (HAPI) refers to the skin and (or) deep tissue injuries of patients 24 hours after admission. PI can cause pain and worsen the prognosis of the disease, and in severe cases, it can cause secondary infection and death. At the same time, it will prolong the hospitalization time, occupy a lot of medical resources and increase the family financial burden. Critically ill patients are always at high risk of PI in medical institutions, and its incidence rate is 3.8 times that of non-critically ill patients. Many risk factors increase the susceptibility of critically ill patients to PI, such as insufficient blood perfusion, low blood oxygen saturation, use of vasoactive drugs, mechanical ventilation or renal replacement therapy. The prevalence of PI in critical patients abroad is 16.9%~23.8%; The prevalence of PI in critically ill patients in China is 5.58% ~ 11.09%; In 2021, Sonia et al. conducted an international multi-center large sample survey (from 1117 intensive care units and 90 countries/regions), and the prevalence of PI in critically ill patients was 16.2%. As we all know, PI is a common chronic refractory wound in clinic, with low cure rate and high treatment cost. Sun Xiaofang followed up 59 PI patients and found that the wound healing time of stage 3 and above PI was about 37 months, and only 5.1% of the patients' wounds were completely healed, with an average cost of about 6,600 yuan. In 2019, the US spent as much as $2.08 billion on PI for critically ill patients. PI is also an important reason for the increase of mortality in critically ill patients. As some critically ill patients are complicated with multiple organ failure, once PI occurs, it is easier to delay infection and cause sepsis, leading to the death of patients. Therefore, how to avoid PI in critically ill patients is the primary problem faced by medical workers.

1.2 PI Risk Assessment Tool for Critically Ill Patients Over the years, it has become a global consensus that prevention of PI is more important than treatment. Risk assessment is the first step to prevent PI, and the accuracy of its results will directly affect the selection of preventive measures and preventive effects. At present, there are Braden scale, Norton scale and Waterlow scale, which are widely used in clinical practice. Norton scale and Waterlow scale are proved to have the best prediction effect in evaluating elderly patients and surgical patients. However, when Braden scale is applied to PI risk assessment of critically ill patients, its predictive ability is moderate (good sensitivity and low specificity), which leads to the implementation of many non-targeted preventive measures in clinic and wastes medical resources. As early as 1990s, foreign scholars compiled PI risk assessment forms for critical patients, including Cubbin &Jackson, SunderLand, SS(Suriadi and Sanada Scale) and EVARUCI. Ye Tong et al. analyzed the reasons why these scales can't be widely used. They are compiled according to the characteristics of foreign critical patients, and some items are not applicable to Chinese population. Secondly, some items need to be calculated before filling in (such as the range of blood pressure drop), and the steps are complicated, which increases the workload of medical staff. Some items are subjective indicators, and the scores of the same patient are quite different, so the ability requirements of evaluators are strict. At present, there is no special PI evaluation scale for critically ill patients based on the characteristics of Chinese population. Generally speaking, the traditional evaluation tools, the evaluation process consumes a lot of manpower, and the items of the scale also greatly affect the accuracy of the evaluation.

In 2019, Sheng Han et al. collected the data of 278 ICU patients by retrospective case-control method, and obtained independent risk factors of stress injury by multivariate analysis: age, edema, hemiplegia, diabetes, acute physiological and chronic health score II, incontinence, and established a nomogram model of stress injury. The area under ROC curve of this model is 0.83, which has good stability and discrimination. However, this model has a small sample size, lacks external verification, and has a high prediction performance bias. Moreover, diabetes, edema, hemiplegia, incontinence, etc. are all classified variables, which can't really quantify the relationship between risk factors and stress injuries.

The pathological mechanism of stress injury is complex and dynamic, including internal and external factors. Dana thinks that tissue tolerance is an intermediate variable between internal and external factors, which reflects the tolerance of tissue to pressure and oxygen, and further puts forward the theoretical framework of stress injury prediction model-patient's own factors (age, comorbidity, gender, body index, etc.) and mechanical factors (friction/shear force, mobility, mobility, etc.). In 2019, the Prevention and Treatment of Stress Injury: A Clinical Practice Guide (hereinafter referred to as the "2019 edition of the Clinical Guide for Stress Injury") published by the European Stress Injury Advisory Committee, the American Stress Injury Advisory Committee and the Pan-Pacific Stress Injury Alliance proposed that the risk assessment of patients should be Consider the effects of basic diseases, such as blood perfusion changes caused by diabetes and neuropathy, which will affect the sensitivity and tolerance of skin. Therefore, when evaluating the risk of patients' PI, medical workers should comprehensively consider the patients' basic diseases and various risk factors, and analyze them individually. By analyzing the adverse events of hospital stress injury in the early stage, it is found that when the condition of critical patients changes, medical workers' awareness of PI risk assessment is insufficient, which may be another important reason why critical patients are more prone to PI. How to comprehensively consider all kinds of risk factors faced by critically ill patients and evaluate risks in real time, PI risk prediction model brings new hope to solve a difficult problem.

1.3 the development status of pi risk prediction model Disease risk prediction model has always been a hot spot in medicine. PI risk prediction model refers to a mathematical model with stress injury risk factors as variables and machine learning algorithm to predict the probability of PI. It can quickly, comprehensively and accurately screen out high-risk patients with PI, and at the same time provide controllable indicators for medical workers, further promote the implementation of targeted treatment and nursing measures, reduce the incidence of PI, and reduce medical expenses.

The clinical data of 486 ICU patients in Deng Xiaohong were collected, and the PI risk prediction model was constructed by using classification regression tree algorithm. The decision tree model consisted of 4 layers and 11 nodes, and three high-risk groups were selected: (1) Age > 81 years old; (2) Age ≤8l, with fecal incontinence; (3) Patients with age ≤81 years old, no fecal incontinence, Braden score ≤13, and diastolic blood pressure < 60 mmHg, the area under the ROC curve of this model is 0.82. There is no internal verification in this study, and the prediction performance of the model may be too high. The selection of PI risk factors in this study is based on literature review rather than evidence-based, and it cannot be determined that risk factors are highly correlated with stress injury.

Yu et al. collected the clinical data of inpatients in 2014-2016, took the results of multi-factor analysis as model prediction variables, and used decision tree, logistic regression and random forest machine learning algorithm to build prediction models to evaluate the risk of PI among inpatients. The results showed that the random forest model had the best prediction performance, and the area under ROC curve was 0.84.

In both studies, a single machine learning algorithm is used to build a stress injury risk prediction model. The life cycle of machine learning is a process of self-learning and using known data sets to build a model to predict the occurrence of unknown data events. First, the best prediction effect can be achieved by selecting an appropriate machine learning algorithm according to the research objective, variable classification and data set attributes. Secondly, whether the missing data can be handled correctly will also affect the prediction performance of the model, because the final effect of the model depends on the amount of data and the amount of useful information contained in the data. Finally, the verification of the model is the most critical. Internal verification can prevent the model from over-fitting, so as to obtain a more reliable and accurate evaluation value. External verification mainly evaluates the prediction performance of the model through clinical application, and analyzes and optimizes the model by using newly collected data, so that the model can be continuously updated dynamically, which provides a basis for the future wide-range use of the model. In this study, the leading artificial energy intelligent models in the world are used to form an algorithm library. Based on the standard data established in the early stage of the project, multiple models in the model library are trained by random and repeated sampling, and the best integrated prediction model is mined. Artificial intelligence model is an integrated learning model (it is a big category of machine learning, which is different from single machine learning model). It completes learning tasks by building multiple learners, mainly including single model training and multi-model fusion. Ensemble learning can fully make up for the deficiency of single machine learning algorithm, and its main advantages are as follows: (1) There is no limit to the types of sub-learners, and the integrated total learners can be homogeneous (same type of sub-learners) or heterogeneous (different types of sub-learners), which improves the performance and compatibility of ensemble learning; (2) Generally, the generalization performance can be significantly superior to that of a single learner through integration. If the sub-learner is weak, this superiority will be even more obvious. PI artificial intelligence model mainly transforms clinical data through six steps: data extraction and cleaning, data set formation, model training, model evaluation and verification, model interpretation and formation of clinical decision information, which will make full use of the useful information in the data. This study will summarize the risk factors of stress injury in critical patients through evidence-based medicine and expert correspondence, and make use of the advantages of integrated learning model to establish a PI artificial intelligence prediction model to ensure its high prediction performance.

1.4 PI artificial intelligence model's clinical application prospect In 2020, the Notice of Further Strengthening Nursing Work in Medical Institutions issued by the National Health and Health Commission pointed out that it is necessary to further promote the development of nursing informatization, promote the deep integration of information technology and nursing work, and establish a nursing management platform with different functions. With the continuous development of information technology, the application of machine learning algorithms to collect and utilize big data has become a development trend. Machine learning algorithm is the core of artificial intelligence. In PI management, by building a PI risk prediction model, not only It can evaluate the PI risk of critically ill patients, realize automatic data analysis and promote the development of PI electronic information management. Park et al. used retrospective research method to collect clinical data of 14,907 inpatients with electronic medical record database, and established cox risk regression model to predict patients' PI risk. The area under ROC curve of this model is 0.95, and its prediction effect is much better than that of Braden scale (area under ROC curve is 0.82). The electronic medical record system contains a lot of patient information (personal information of patients, medical records, test results, medication information, etc.). The PI artificial intelligence prediction model is embedded in the electronic medical record system, which can transform the patient's records and data into valuable medical information. It is expected to provide a new direction for early prevention, continuously monitor the risk of patients' stress injury, and promote medical workers to introduce effective treatment and care. It can provide appropriate medical advice for patients and their families, facilitate the implementation of clinical decision-making based on evidence, and ultimately reduce the occurrence of stress injuries in critically ill patients, improve nursing quality and reduce medical expenses.It can evaluate the PI risk of critically ill patients, realize automatic data analysis and promote the development of PI electronic information management. Park et al. used retrospective research method to collect clinical data of 14,907 inpatients with electronic medical record database, and established cox risk regression model to predict patients' PI risk. The area under ROC curve of this model is 0.95, and its prediction effect is much better than that of Braden scale (area under ROC curve is 0.82). The electronic medical record system contains a lot of patient information (personal information of patients, medical records, test results, medication information, etc.). The PI artificial intelligence prediction model is embedded in the electronic medical record system, which can transform the patient's records and data into valuable medical information. It is expected to provide a new direction for early prevention, continuously monitor the risk of patients' stress injury, and promote medical workers to introduce effective treatment and care. It can provide appropriate medical advice for patients and their families, facilitate the implementation of clinical decision-making based on evidence, and ultimately reduce the occurrence of stress injuries in critically ill patients, improve nursing quality and reduce medical expenses.

ELIGIBILITY:
Inclusion Criteria:

* Length of ICU stay > 48 h
* Be at least 18 years old
* Meet the diagnostic criteria of intensive care unit and APACH II <35 points

Exclusion Criteria:

* Patients with skin diseases and burns
* Patients with pressury injury at admission
* Repeat hospitalization
* Died 24 hours after pressure injury.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients This study was a retrospective study, and all patients meeting the admission criteria were selected from the Intensive Care Unit (ICU) of a tertiary comprehensive university-affiliated hospital from January 2016 to December 2021 (34 beds were provided for critical care, and 2,686 patients were admitted during the study period).
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Hospital-acquired pressure injury | 2023-03-01
  The staging assessment of pressure injuries was based on the 2016 edition of the American Pressure Injury Expert Advisory Group Guidelines(WOCN 2016 Guideline).

CONTACTS AND LOCATIONS:
Overall Officials: YangChaonan Nurse-in-charge, BM, Study Chair — Huzhou University

IPD SHARING:
Plan to Share IPD: Undecided
The research has not yet been carried out. It is expected that the data will be collected in October and the pressure injury risk prediction model will be established. After seeing the effect of the model, the team will decide whether to open the patient data or not.

REFERENCES:
- [Result] Gaspar S, Botelho Guedes F, Vitoriano Budri AM, Ferreira C, Gaspar de Matos M. Hospital-acquired pressure ulcers prevention: What is needed for patient safety? The perceptions of nurse stakeholders. Scand J Caring Sci. 2022 Dec;36(4):978-987. doi: 10.1111/scs.12995. Epub 2021 Jun 9. PMID 34105825
- [Result] Stotts NA, Brown DS, Donaldson NE, Aydin C, Fridman M. Eliminating hospital-acquired pressure ulcers: within our reach. Adv Skin Wound Care. 2013 Jan;26(1):13-8. doi: 10.1097/01.ASW.0000425935.94874.41. PMID 23263395
- [Result] Spruce L. Strategies to Help Prevent Hospital-Acquired Pressure Injuries. AORN J. 2020 Feb;111(2):241-242. doi: 10.1002/aorn.12952. No abstract available. PMID 31997318
- [Result] Wood J, Brown B, Bartley A, Margarida Batista Custodio Cavaco A, Roberts AP, Santon K, Cook S. Reducing pressure ulcers across multiple care settings using a collaborative approach. BMJ Open Qual. 2019 Aug 20;8(3):e000409. doi: 10.1136/bmjoq-2018-000409. eCollection 2019. PMID 31523723
- [Result] Krupp AE, Monfre J. Pressure ulcers in the ICU patient: an update on prevention and treatment. Curr Infect Dis Rep. 2015 Mar;17(3):468. doi: 10.1007/s11908-015-0468-7. PMID 25821191
- [Result] Coyer F, Miles S, Gosley S, Fulbrook P, Sketcher-Baker K, Cook JL, Whitmore J. Pressure injury prevalence in intensive care versus non-intensive care patients: A state-wide comparison. Aust Crit Care. 2017 Sep;30(5):244-250. doi: 10.1016/j.aucc.2016.12.003. Epub 2017 Jan 4. PMID 28063724
- [Result] Lima Serrano M, Gonzalez Mendez MI, Carrasco Cebollero FM, Lima Rodriguez JS. Risk factors for pressure ulcer development in Intensive Care Units: A systematic review. Med Intensiva. 2017 Aug-Sep;41(6):339-346. doi: 10.1016/j.medin.2016.09.003. Epub 2016 Oct 22. English, Spanish. PMID 27780589
- [Derived] Chaonan Y, Ji C, Huibin P, Shen L, Xiaohong L. Risk Factors for Pressure Injury in ICU Patients. Nurs Open. 2026 Feb;13(2):e70384. doi: 10.1002/nop2.70384. PMID 41618576